CLINICAL TRIAL: NCT01196468
Title: HIV Indicator Diseases Survey Across Europe
Brief Title: HIV Indicator Diseases Survey Across Europe - UK Arm
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Collaborators: HIV in Europe (Co-Sponsor) (Unknown)
Responsible Party: Dr Ann Sullivan, Chelsea and Westminster NHS Foundation Trust, London, UK
Other Study IDs: Indicator Diseases Survey
Record Dates: First submitted 2010-08-10; First posted 2010-09-08 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2009-10

CONDITIONS: HIV; AIDS; Indicator Diseases/Indicator Conditions
Keywords: HIV; Testing; Targeted; Indicator; Diseases; Anal dysplasia; Cervical dysplasia; STI; Lymphoma; Seborrhoeic dermatitis; Exanthema; Thrombocytpaenia; Lymphopaenia; Hypergammaglobulinaemia
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Disease; Uterine Cervical Dysplasia; Sexually Transmitted Diseases; Lymphoma; Dermatitis, Seborrheic; Exanthema; Hypergammaglobulinemia | interventions — HIV Testing; Interviews as Topic

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Salivary or serological HIV test
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Anal/cervical dyplasia: Any patient presenting for care with any degree of anal or cervical dysplasia
  Interventions: Other: HIV test (serological or salivary); Other: Interview
- STI: Any patient presenting for care with any non-HIV sexually transmitted infection
  Interventions: Other: HIV test (serological or salivary); Other: Interview
- Lymphoma: Any patient presenting for care with malignant lymphoma of any histological type
  Interventions: Other: HIV test (serological or salivary); Other: Interview
- Seborrhoeic dermatitis/exanthema: Any patient presenting for care with seborrhoeic dermatitis/exanthema
  Interventions: Other: HIV test (serological or salivary); Other: Interview
- Thromobocytopaenia/Leucopaenia, or hypergammaglobulinaemia: Any patient presenting for care with unexplained thromobocytopaenia/leucopaenia of more than four weeks duration, or with hypergammaglobulinaemia
  Interventions: Other: HIV test (serological or salivary); Other: Interview

INTERVENTIONS:
Other: HIV test (serological or salivary) — An HIV test will be offered to all patients accessing the healthcare setting for care of the "indicator" condition
Other: Interview — Demographic data will be collected for each patient consenting to an HIV test. With informed written consent, additional data will be collected from patients via focussed interview. Data comprises: previous medical history, previous health seeking behaviours, previous HIV testing history, previous viral hepatitis testing/diagnosis history, and assessment of HIV acquisition risk factors

SUMMARY:
In Europe many patients infected with HIV remain undiagnosed, although this percentage varies between 15-80% across the continent. In the UK it is estimated to be 27%. Undiagnosed HIV results in increased morbidity and mortality and reduced treatment response, as appropriate health interventions are delayed. It also has adverse public health implications, with those individuals unaware of their HIV status being more likely to transmit the virus.

An important public health issue is how to diagnose more individuals with HIV earlier in the course of their infection. In the US, the Centre for Disease Control and Prevention (CDC) has introduced testing guidelines whereby all individuals are tested, unless they object, at any point of contact with the healthcare system - the "opt-out" testing guidelines.

At the "HIV in Europe" Conference held in November 2007, the consensus, which included patient and public involvement, was that such an approach would not be suitable for Europe. The Conference recommended further development of focused HIV testing in patients presenting with certain clinical conditions and diseases - the "indicator disease'' testing guidelines.

Cost effectiveness analyses suggests cost savings if a screened population has an HIV prevalence of at least 1%, although this rate may be as low as 0.1%. However, there is very little - if any - evidence regarding HIV prevalence for certain conditions and diseases in specific and easy to identify sections of society. The focus of attention is on those conditions and diseases which occur more frequently in individuals known to be infected with HIV.

The aim of this study is to assess HIV prevalence for several diseases and conditions, within a specific segment of the population not yet diagnosed with HIV, who present for care with that specific disease or condition. These conditions have been selected as they occur frequently in individuals already diagnosed with HIV infection. This is a pilot study to inform phase two, which will involve more diseases and conditions with a wider participation of centres across Europe.

ELIGIBILITY:
Inclusion criteria

* Aged 16 years and over
* Presenting for care with one of the indicator diseases or conditions:

  * A sexually transmitted disease
  * Malignant lymphoma
  * Cervical or anal dysplasia or cancer
  * Unexplained leukocytopenia or thrombocytopenia lasting at least 4 weeks, or hypergammaglobulinaemia
  * Seborrheic dermatitis or exanthema
* sub-study - consents to providing additional information

Exclusion criteria

* Known HIV positive
* sub-study - declines to consent for additional information to be collected

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults (16 years and over), not known already to be HIV-positive, presenting for care in designated healthcare settings with one of five "indicator diseases." Sequential patients will be offered HIV tests, and if they accept, asked to provide additional information via focussed interview (sub-study).
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-07 (Actual); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Prevalence of HIV infection in patients presenting to specific services with specific HIV indicator diseases

SECONDARY OUTCOMES:
Previous HIV testing behaviour of individuals presenting with an indicator disease or condition (sub-study only)
  Any previous history of HIV tests taken: total number, dates, and results
Demographic data of individuals presenting for care with specified indicator diseases
  Data comprise: age group, sex, ethnicity (plus sexuality and injecting drug use history for sub-study participants only)
Time to transfer to care for those individuals testing HIV positive
Immune status of newly-diagnosed HIV positive individuals as determined by CD4 cell count
HIV risk factors (sub-study only)
Previous medical history and health-seeking behaviour (sub-study only)
  Past medical history will be recorded, with particular attention paid to previous illnesses that constitute AIDS-defining illnesses, or other severe, non-AIDS infections and cancers. Number of visits to primary care and any inpatient admissions over preceding five years will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ann K Sullivan, MBBS FRCP, Principal Investigator — Chelsea and Westminster NHS Foundation Trust; Jens Lundgren, MBBS, Study Director — University of Copenhagen and Righospitalet; David Cunningham, PhD FRCP, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Chelsea and Westminster NHS Foundation Trust, London
  - Royal Marsden NHS Foundation Trust, London